CLINICAL TRIAL: NCT06380231
Title: a Randomized Controlled Experimental Design That Uses a Pretest-Posttest Control Group Model.
Brief Title: Skin-to-skin Contact Between Premature Infant and Mother
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Rumeli University (Other)
Responsible Party: Principal Investigator, Yazile Sayin, Researcher, PhD, Istanbul Rumeli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRU-YAZILE-001
Record Dates: First submitted 2024-03-09; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Kangaroo-mother Care
Keywords: premature; kangaroo mother care; heart rate; oxygen saturation; perfusion index
MeSH Terms: conditions — Premature Birth | interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kangaroo mother care (KMC) for experimental group (Experimental): Examined physiological parameters of both groups were measured before, during and after KMC and traditional mother's bosom. This measurement was made at 15-minute intervals for 45 minutes (0-01,15,30,45 minutes). Physiological parameters before and after KMC and traditional mother's bosom represent incubator conditions.
  Interventions: Other: kangaroo mother care (KMC)
- control group (No Intervention): The control group received only traditional mother's bosom. In the control group, unlike the experimental group, the mother's clothes were not removed. The hands of the mothers were cleaned with 0.4% chlorhexidine, and the mothers were seated in the KMC chair. The same chair was used for the experimental and control groups.
  A hospital shirt was placed over the mother's own clothes for hygiene purposes only. The baby was not naked, was given to his mother wrapped in a blanket. The infant spent 45 minutes in traditional mother's bosom without skin-to-skin contact. There were no restrictions placed on the position of the mother holding the infant, and she could hold the infant upright, horizontally, and to the right or left. In control groups, all mothers were permitted to sing lullabies or talk to their infants if they chose to do so.

INTERVENTIONS:
Other: kangaroo mother care (KMC) — Kangaroo mother care is a simple care that aims to protect the health and well-being of premature babies, where skin-to-skin contact is achieved by placing the premature baby in an upright position, face down, between the parent's breasts, wearing only a diaper and a cap.
  Before the experimental group infant was given to the mother, his/her hat was put on, and clothes were removed. The infant was placed in an upright position (approximately 60°) between the mother's two breasts. To enable the infant to breathe, his/her head was positioned to the right or left with ear touching the mother's chest, arms and legs were flexed, and hip was abducted. The mother supported the infant's neck and back with one hand and the hips with the other. The infant's back was covered with a cotton blanket. An noninvasive pulse Co-oximetry was attached to the right wrist of the infant to evaluate heart rate, oxygen saturation, and perfusion index.
  Arms: kangaroo mother care (KMC) for experimental group

SUMMARY:
Aim: To determine the effect of kangaroo mother care (KMC) on perfusion index, heart rate, and oxygen saturation in premature infants who were discharged early and admitted to the neonatal intensive care in the following days.

DETAILED DESCRIPTION:
METHOD Design: This study has a randomized controlled experimental design and uses a pretest-posttest control group model. Consolidated Standards of Reporting Trials (CONSORT) guidelines were followed throughout the study protocol.

Experimental (n = 38) and control (n = 38) groups were assigned using the simple randomization technique at the neonatal intensive care unit (NICU) of private an university hospital in Istanbul, Turkey. Heart rate, perfusion index and oxygen saturation levels of the experimental group in which KMC was applied and the control group in which KMC was not applied were compared. Data were collected via the Mother and Infant Introductory Information Form, Kangaroo Mother Care Preparation Checklist, Kangaroo-Mother Care- Physiological Parameter Monitoring Form, and Noninvasive Pulse Co-Oximetry.

Setting: The study was conducted on premature infants receiving incubator care in the NICU of a private university hospital in Istanbul, Turkey. There are 15 nurses (one of whom is the charge nurse), one neonatologist, three assistant doctors, five auxiliary staff members, and one secretary working in the NICU. The research nurse in this study also worked in the NICU where the study was conducted.

The NICU has a bed capacity of 10 and15 and contains 20 incubators with monitors, six mechanical ventilators, nine vital monitoring devices, one isolation, one milk and formula preparation, one medication preparation, and one lactation station. There is a special section in the breastfeeding room, reserved for KMC, with a fully equipped incubator and monitor. The KMC room has a chair, an incubator and a monitor which have noninvasive pulse co-oximetry (NIS-pulse co-oximeter).

KMC is a doctor's order for babies hospitalized in NICU and is applied routinely. If you don't mind, the doctor recommends KMC to all babies twice a day. It was only applied once a day during the Coronavirus-19 pandemic period.

Data Collection Tools: In this study, three forms and noninvasive pulse co-oximetry (MR NI-pulse co-oximeter) were used to collect data. Mother and Baby Identification Information Form (MIIF) includes the mother's age, social security, smoking and alcohol history and history, gender, birth, birth cycle positive ventilation status, postnatal APGAR score, gestational age and weight. This form was prepared from patient files and literature information.

The Kangaroo Mother Care Preparation Checklist (KMCPC) is a list of mother and baby's preparation for KMC. The form includes information such as clothing, hygiene, position, duration, temperature protection for mother and baby and was developed in accordance with the literature.

Kangaroo-Mother Care-Physiological Parameter Monitoring Form (KMC-PPMF) is a form in which information about the baby's perfusion index, heart rate and premature oxygen saturation is recorded during, before and after the KMC. KMC-PPMF is a form prepared and used by the Research and Application Hospital Quality Unit and the Cronbach alpha value of the form is 0.777 (good level).

MR NIS-pulse co-oximeter has been used in all intensive care units in recent years. MR NIS-pulse co-oximeter have a spectrophotometric sensor that may be an adhesive single use for continuous monitoring or a reusable finger clip sensor for spot check assessments. It has been reported that noninvasive hemoglobin (Hb) monitoring with pulse CO-oximetry may be useful in the early detection of Hb changes in newborns. MR noninvasive spectrophotometric (NIS)-pulse co-oximeter is a noninvasive monitoring device featuring pulse oximetry with the option to measure multiple additional parameters: such as perfusion index, heart rate and oxygen saturation, total hemoglobin, respiration rate.

Mother-Infant Preparation and KMC: The KMC is a separate section with an incubator inside the breastfeeding room in the NICU. The space was kept at a temperature of 24 and 26°C, was private, and had no air circulation and little noise or light. The room contained a clean hospital shirt for mothers to wear when they removed their top clothes and a seat where they could sit comfortably with their infants. To minimize fluctuations in KMC biorhythms, measurements were recorded at the same time every 24-hour for both the experimental and control groups.

All mothers were instructed to take a bath before coming to the hospital and not to wear perfume, body cream, accessories, or makeup.

Experimental Group: The purpose of the study was explained to the mothers of the experimental group infants selected for the study by the researcher nurse, written informed consent was obtained, KMC was explained and demonstrated to the mothers, and an illustrated NICU brochure was given to them for review. The easiest part of this research was that the vast majority of mothers were knowledgeable about KMC because it was already practiced in the NICU. The mothers only requested additional details about information related to wearing jewelry, perfume, or lotion.

On the day of KMC, the experimental group mother was taken to the KMC room, her upper garment was removed, and a clean front-opening hospital shirt was put on. The hands, abdomen, and breasts of the mothers were cleaned with 0.4% chlorhexidine, and the mothers were seated in the KMC chair. All infants were fed and their diapers changed one hour before being handed over to their mothers. The mothers were made to warm their hands by rubbing them before holding the infant in their hands.

The Control Group: The control group don't received KMC.

Statistical Analysis: To examine the distribution of the data, skewness and kurtosis values were examined with the Shapiro-Wilk-Kolmogorov-Smirnov test (p>0.005). According to the Kolmogorov-Smirnov test, the data were normally or nearly normally distributed between -2/+2 (p>0.005). While Pearson correlation coefficient (r) was used to analyze the relationships between normal data, frequency and percentage (N and %), mean and standard deviation (Mean ± SD), Chi-square test (χ2), Fisher exact test and independent sample t-test were used in the analysis of qualitative and quantitative variable data. The Statistical Package for Social Sciences, version 22.0 software (IBM Corp.; Armonk, New York, USA) was used. The p-values lower than 0.05 were considered statistically significant.

The data on the physiological parameters (perfusion index, heart rate and oxygen saturation) of experimental and control group babies were in vivo measurements. The deviations of these data from the arithmetic mean were shown as mean and standard deviation. Statistics of these data were performed with the independent sample t-test. Pearson's chi-square test was used to determine the relationship between categorical data such as mode of delivery, status of receiving positive pressure ventilation, and reason for NICU admission were analysed using. Since the expected values related to mode of delivery and gender were low, Fisher's Exact test was used.

Random Block Scheme: Although the homogeneity of the groups was tried to be preserved in the study with sampling criteria and unbiased assignment, the similarity and effects of the variables cannot be guaranteed. In this case, the random block order was important. The block design could be applied to the control group. After collecting the data of the control group babies, the researcher performed KMC on these babies upon the doctor's request within two hours and recorded the physiological parameters. Under these conditions, the effect of KMC was similar in both the experimental and the control group where the random block was applied, and the difference was statistically insignificant. Significance values of 0, 15 th, 30 th and 45 th minutes regarding perfusion index, peak heart rate and oxygen saturation of the experimental and control groups in a random block scheme: (Equal variances assumed, p = 0.328, p = 0.058, p = 0.132 for 0 th minutes, p = 094, p = 0.091, p = 0.292 for 15 th minutes, p = 0.064 p = 0.108, p =0.060 for 30 th minutes, p = 0.066 p = 0.202, p = 0.245 for 45 th minutes). The experimental and control groups are homogeneous and have similar results during KMC.

ELIGIBILITY:
Inclusion Criteria:

* Baby inclusion criteria: Babies should be admitted to NICU after early discharge, their gestational age should be between 24-37 weeks, the reason for admission to the intensive care unit should be stabilized by the doctor,

Mother inclusion criteria: mother's consent for research, and experimental group mothers' compliance with the dressing rules for KMC, mothers with premature infants who were born at the facility and admitted to the NICU for care were eligible to participate in the present study. Mothers with babies who are discharged early because they are considered medically stable as determined.

Exclusion Criteria:

* Baby exclusion criteria: Congenital anomaly, hemodynamic instability, hydrocephalus, encephalopathy, genetic malformations, chromosomal syndromes, requiring respiratory support, apnea and bradycardia, a skin disorder causing loss of body heat, arterial or intravenous catheter blocking KMC, corticosteroids and sedation treatment.

Mother exclusion criteria: being under 18 years old, cesarean section, mentally and spiritually unhealthy, with skin diseases.

Ages: 24 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
power analysis | two months
  For the sample size, we considered Cohen "s effect size (d) value, which is the acceptable limit in the field of health sciences.
  The sample size was calculated by a t-test in the G*Power 3.1.7 program.

SECONDARY OUTCOMES:
The effect of kangaroo mother care | Examined physiological parameters of both groups were measured before, during and after KMC and traditional mother's bosom . This measurement was made at 15-minute intervals for 45 minutes (0-01th,15th,30th,45 th minutes)
  Perfusion index, heart rate and oxygen saturation were monitored with noninvasive pulse co-oximetry. Examined these physiological parameters of experimental and control groups were measured before and after KMC and traditional mother's bosom (TMB). This measurement was made at 15-minute intervals for 45 minutes (0-01 th ,15 th ,30 th ,45 th minutes). Physiological parameters before and after KMC and TMB represent incubator conditions.
  Data about the baby and the mother were collected with the Mother and Baby Identification Information Form: the mother's age, social security, smoking and alcohol history and history, gender, birth, birth cycle positive ventilation status, and the baby's postnatal activity, pulse, grimace, appearance, and respiration score, gestational age and kilo in weight.
  The preparation of mother and baby for kangaroo mother care were done with The Kangaroo Mother Care Preparation Checklist.

CONTACTS AND LOCATIONS:
Locations (1):
- TC Istanbul Rumeli University, Istanbul, Haliç, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
After the research is accepted for publication, participant data, Study Protocol, Statistical Analysis Plan, Informed Consent Form, Clinical Study Report will be shared.

REFERENCES:
- [Background] George, D., & Mallery, M. (2010).SPSS for windows step by step: A simple guide and reference, 17.0 update (10a ed.) Boston: Pearson
- [Background] Karaagaoglu, E. (2013). An experimental design technique: Randomized block design. Turkish Journal of Biochemistry, 38 (1): 1-4
- [Background] Nyqvist KH; Expert Group of the International Network on Kangaroo Mother Care; Anderson GC, Bergman N, Cattaneo A, Charpak N, Davanzo R, Ewald U, Ludington-Hoe S, Mendoza S, Pallas-Allonso C, Pelaez JG, Sizun J, Widstrom AM. State of the art and recommendations. Kangaroo mother care: application in a high-tech environment. Acta Paediatr. 2010 Jun;99(6):812-9. doi: 10.1111/j.1651-2227.2010.01794.x. Epub 2010 Mar 8. PMID 20219028
- [Background] Cristobal Canadas D, Bonillo Perales A, Galera Martinez R, Casado-Belmonte MDP, Parron Carreno T. Effects of Kangaroo Mother Care in the NICU on the Physiological Stress Parameters of Premature Infants: A Meta-Analysis of RCTs. Int J Environ Res Public Health. 2022 Jan 5;19(1):583. doi: 10.3390/ijerph19010583. PMID 35010848
- [Background] Kommers DR, Joshi R, van Pul C, Atallah L, Feijs L, Oei G, Bambang Oetomo S, Andriessen P. Features of Heart Rate Variability Capture Regulatory Changes During Kangaroo Care in Preterm Infants. J Pediatr. 2017 Mar;182:92-98.e1. doi: 10.1016/j.jpeds.2016.11.059. Epub 2016 Dec 15. PMID 27989406
- [Background] Lee J, Parikka V, Lehtonen L, Soukka H. Parent-infant skin-to-skin contact reduces the electrical activity of the diaphragm and stabilizes respiratory function in preterm infants. Pediatr Res. 2022 Apr;91(5):1163-1167. doi: 10.1038/s41390-021-01607-2. Epub 2021 Jun 4. PMID 34088986
- [Background] Pados BF, Hess F. Systematic Review of the Effects of Skin-to-Skin Care on Short-Term Physiologic Stress Outcomes in Preterm Infants in the Neonatal Intensive Care Unit. Adv Neonatal Care. 2020 Feb;20(1):48-58. doi: 10.1097/ANC.0000000000000596. PMID 30893092
- [Background] Jamal, A.Z., & John, B.M. (2020). Efficacy of noninvasive hemoglobin measurement by pulse co-oximetry in neonates. J Clin Neonatol., 9:57-62. Doi 10.4103/jcn.JCN_89_19
- [Background] Nicholas C, George R, Sardesai S, Durand M, Ramanathan R, Cayabyab R. Validation of noninvasive hemoglobin measurement by pulse co-oximeter in newborn infants. J Perinatol. 2015 Aug;35(8):617-20. doi: 10.1038/jp.2015.12. Epub 2015 Mar 5. PMID 25742288
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343